CLINICAL TRIAL: NCT02492360
Title: Establishing of Neuronal-like Cells From Patients With Cisplatin-Induced Peripheral Neuropathy
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Costantine Albany (Other)
Responsible Party: Sponsor-Investigator, Costantine Albany, Clinical Faculty, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: IRB #1504498959 (IUSCC-0516)
Record Dates: First submitted 2015-05-13; First posted 2015-07-08 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Nervous System Diseases; Testicular Neoplasms
Keywords: Peripheral Neuropathies; Testicular Cancer; Cisplatin; Pharmacogenomics
MeSH Terms: conditions — Peripheral Nervous System Diseases; Testicular Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be obtained from all patients so that peripheral blood mononuclear cells (PBMCs) can be isolated and stored for the eventual creation of iPS cells. iPS cells have the potential to make human neurons that the researchers would like to use for functional studies of specific genes/genetic variants. All samples will also be tested for infectious diseases (Hepatitis B, Hepatitis C, HIV 1 and HIV 2).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Severe Toxicity Group: Diagnosis of testicular cancer; History of any grade 3 or higher peripheral neuropathy after receiving standard dose cisplatin completed more than 1 year but within the last 5 years; Long-term persistence (> 6 months) of grade 2 or higher peripheral neuropathy after completion of a cisplatin containing regimen. Interventions: blood sample collection and report of peripheral neuropathy after cisplatin therapy.
  Interventions: Procedure: Blood sample collection; Behavioral: Report of peripheral neuropathy after cisplatin therapy
- Control Group: Diagnosis of testicular cancer; No history of neurotoxicity (grade 0-1) after completion of a standard cisplatin-containing chemotherapy regimen completed more than 1 year but within the last 5 years; Matched to a specified subject with neurotoxicity based on age (within 10 years), chemotherapy regimen or total cisplatin dosage. Interventions: blood sample collection and report of peripheral neuropathy after cisplatin therapy.
  Interventions: Procedure: Blood sample collection; Behavioral: Report of peripheral neuropathy after cisplatin therapy

INTERVENTIONS:
Procedure: Blood sample collection — Six tubes of blood will be collected during one blood draw.
Behavioral: Report of peripheral neuropathy after cisplatin therapy — Twenty questions about the peripheral neuropathy the patient is currently experiencing, and twenty questions about the worst peripheral neuropathy the patient ever experienced after cisplatin treatment.

SUMMARY:
This study targets patients with cisplatin-induced peripheral neuropathy and will allow us to: a) study peripheral neuropathy in diverse human sensory neurons in ways that were not possible previously; b) gain insight on druggable targets to treat or prevent this devastating side effect of chemotherapy; c) provide a human cellular model that can be used for screening of drugs to determine if they are neurotoxic. The combination of patient information and in vitro measurements provides a highly relevant and clinically useful model for studies aimed to impact treatment selection for the individual cancer patient.

DETAILED DESCRIPTION:
Primary Objective-To establish a biobank of specimens that allows for the future creation of iPS cells with the potential to make human neurons for functional studies of specific genes/genetic variants.

Secondary Objectives-To develop a clinically relevant in vitro model of cisplatin induced peripheral neuropathy to be used to 1) screen new drugs for the treatment or prevention of peripheral neuropathy; 2) evaluate candidate genes for their role in cisplatin induced neuropathy.

Study Procedures-Subjects who wish to participate will undergo the following study procedures, which will be performed after the informed consent document is obtained:

1. Sample Collection-A trained phlebotomist will conduct a blood draw for the collection of SIX samples for peripheral blood mononuclear cell (PBMC) isolation and infectious disease testing.
2. Patient Self-Report of Toxicities-All patients in the study will be asked to fill out the Patient-reported Toxicity Form. This will take approximately 10 minutes to complete and consists of 20 questions related to patient symptoms describing toxicities experienced secondary to receiving cisplatin chemotherapy. They will be asked to fill out the form twice: (1) describing the peripheral neuropathy they currently are experiencing and (2) describing the worst peripheral neuropathy toxicity they experienced as a result of cisplatin therapy. These paper forms will be filled out at time of enrollment in the study.
3. Physician Report of Toxicities-The patient's physician or the designatee will complete an adverse event form at day of enrollment detailing the physician's assigned grade of toxicities (according to CTCAE version 4.3) experienced from cisplatin. Other information regarding the particularly severe neurotoxicity may also be collected from physicians (e.g. patient use of walker or wheelchair, patient application for disability based on neuropathy).
4. General Information- This information will be collected at the same time point as all of the other study procedures (i.e., Day One). This will include but may not be limited to: age, height, weight, patient-identified race and ethnicity, information about the chemotherapy regimen, total cisplatin dose administered and date of last cisplatin dose.
5. Cisplatin Dose-Total cumulative dose of cisplatin administered will be recorded. Outside records will be obtained where needed.
6. Follow-up and Duration of Follow-Up-There will be no subsequent patient follow-up after time of enrollment. Subjects may withdraw consent for specimen use by contacting the PI in writing.

ELIGIBILITY:
Inclusion Criteria---Severe Toxicity Group

1. Diagnosis of testicular cancer
2. Age ≥ 18 years at the time of informed consent
3. Male
4. History of any grade 3 or higher peripheral neuropathy after receiving standard dose cisplatin completed more than 1 year but within the last 5 years
5. Long-term persistence (> 6 months) of grade 2 or higher peripheral neuropathy after completion of a cisplatin containing regimen.
6. Patient understands the nature of the study and provides written informed consent

Inclusion Criteria---Control Group

1. Diagnosis of testicular cancer
2. Age ≥ 18 years
3. Male
4. No history of neurotoxicity (grade 0-1) after completion of a standard cisplatin-containing chemotherapy regimen completed more than 1 year but within the last 5 years
5. Matched to a specified subject with neurotoxicity based on age (within 10 years), chemotherapy regimen or total cisplatin dosage
6. Patient understands the nature of the study and provides informed consent

Exclusion Criteria (Both groups)

1. Treatment with other severely neurotoxic chemotherapy prior to or concomitantly with cisplatin.
2. Presence of peripheral neuropathy prior to cisplatin therapy
3. Poorly controlled or insulin-dependent diabetes or other conditions likely to predispose neurotoxicity (alcoholism, Charcot-Marie-Tooth disease)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of two groups: testicular cancer patients with severe neuropathy (experimental group) and testicular cancer patients without neuropathy (control group). One control subject will be recruited for each experimental subject with severe neurotoxicity. Controls will be matched based on age (within 10 years), tumor type, race, ethnicity, and chemotherapy regimen and cumulative dose of cisplatin during which the toxicity occurred.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Biobank of peripheral blood mononuclear cells (PBMCs) | Once (at enrollment)
  PBMCs will be used for the future creation of iPS cells with the potential to make human neurons

CONTACTS AND LOCATIONS:
Overall Officials: Costantine Albany, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Simon Cancer Center, Indianapolis, Indiana, United States